CLINICAL TRIAL: NCT02044653
Title: Phase II Clinical Trial to Explore the Optimal Fixed Starting Dose & Dosing Interval and to Evaluate the Safety of GX-E2 in the Anemic Patients Diagnosed With Chronic Kidney Disease and Receiving Hemodialysis (HD) / Peritoneal Dialysis (PD)
Brief Title: Study to Evaluate the Efficacy and Safety of GX-E2 in the Anemic Patients Diagnosed With Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GX-E2_P2
Record Dates: First submitted 2014-01-09; First posted 2014-01-24 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Anemia; Chronic Kidney Disease
Keywords: Phase 2
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GC1113; Darbepoetin alfa; continuous erythropoietin receptor activator

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- Group A (Part A) (Experimental): GX-E2 : Subcutaneously injection every 2 weeks (Q2W) at dose 3ug/kg
  Interventions: Drug: GX-E2
- Group B (Part A) (Experimental): GX-E2 : Subcutaneously injection every 2 weeks (Q2W) at dose 5ug/kg
  Interventions: Drug: GX-E2
- Group C (Part A) (Experimental): GX-E2 : Subcutaneously injection every 2 weeks (Q2W) at dose 8ug/kg
  Interventions: Drug: GX-E2
- Group D (Part A) (Experimental): GX-E2 : Subcutaneously injection every 4 weeks (Q4W) at dose 3ug/kg
  Interventions: Drug: GX-E2
- Group E (Part A) (Experimental): GX-E2 : Subcutaneously injection every 4 weeks (Q4W) at dose 5ug/kg
  Interventions: Drug: GX-E2
- Group F (Part A) (Experimental): GX-E2 : Subcutaneously injection every 4 weeks (Q4W) at dose 8ug/kg
  Interventions: Drug: GX-E2
- Group G (Part B) (Experimental): GX-E2 : Subcutaneously injection every 2 weeks (Q2W) at dose 5ug/kg
  Interventions: Drug: GX-E2
- Group H (Part B) (Experimental): GX-E2 : Subcutaneously injection every 2 weeks (Q2W) at dose 8ug/kg
  Interventions: Drug: GX-E2
- Group I (Part B) (Active Comparator): MIRCERA : Subcutaneously injection every 2 weeks (Q2W) at dose 0.6ug/kg
  Interventions: Drug: MIRCERA
- Group J (Part B) (Experimental): GX-E2 : Intravenously injection every week (Q1W) at dose 5ug/kg
  Interventions: Drug: GX-E2
- Group K (Part B) (Experimental): GX-E2 : Intravenously injection every week (Q1W) at dose 8ug/kg
  Interventions: Drug: GX-E2
- Group L (Part B) (Experimental): GX-E2 : Intravenously injection every 2 weeks (Q2W) at dose 8ug/kg
  Interventions: Drug: GX-E2
- Group M (Part B) (Active Comparator): NESP : Intravenously injection every week (Q1W) at dose 30ug
  Interventions: Drug: NESP

INTERVENTIONS:
Drug: GX-E2 — Each Group of Peritoneal dialysis patients (n=10) will be administered GX-E2 3ug/kg to 8ug/kg
  Other Names: GC1113
  Arms: Group A (Part A); Group B (Part A); Group C (Part A); Group D (Part A); Group E (Part A); Group F (Part A)
Drug: GX-E2 — Each Group of Peritoneal dialysis patients (n=24) will be administered GX-E2 5ug/kg to 8ug/kg
  Other Names: GC1113
  Arms: Group G (Part B); Group H (Part B)
Drug: GX-E2 — Each Group of Hemodialysis patients (n=30) will be administered GX-E2 5ug/kg to 8ug/kg
  Other Names: GC1113
  Arms: Group J (Part B); Group K (Part B); Group L (Part B)
Drug: NESP — Each Group of Hemodialysis (n=30) will be administered NESP 30ug
  Other Names: Aranesp; Darbepoetin alfa
  Arms: Group M (Part B)
Drug: MIRCERA — Each Group of Peritoneal dialysis (n=24) will be administered MIRCERA 0.6ug/kg
  Other Names: Methoxy Polyethylene glycol-epoetin beta
  Arms: Group I (Part B)

SUMMARY:
The primary objective of study is

* Part A : To explore the optimal fixed starting dose and dosing interval of GX-E2
* Part B : To evaluate the proof of concept (POC) of GX-E2

DETAILED DESCRIPTION:
The secondary objective of study is to evaluate:

* change of red blood cell indices in anemic patients with chronic kidney disease receiving hemodialysis/peritoneal dialysis when administering GX-E2 intravenously/subcutaneously
* change of reticulocyte indices in anemic patients with chronic kidney disease receiving hemodialysis/peritoneal dialysis when administering GX-E2 intravenously/subcutaneously
* safety of GX-E2 when administering intravenously/subcutaneously
* incidence of blood transfusion in anemic patients with chronic kidney disease receiving hemodialysis/peritoneal dialysis when administering GX-E2 intravenously/subcutaneously
* Immunogenicity in anemic patients with chronic kidney disease receiving hemodialysis/peritoneal dialysis when administering GX-E2 intravenously/subcutaneously

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ≥18 yr of age
* Chronic Kidney diseases with hemodialysis, peritoneal dialysis with Kt/V ≥ 1.2 (hemodialysis) or Kt/V ≥ 1.7 (peritoneal dialysis) within a year
* Adequate transferrin saturation (≥20%), serum ferritin (≥100ug/L)
* Should have received Vitamine B12 ≥ 3 months before the first dose of study agent
* Should have received Folate ≥3 months before the first dose of study agent
* No erythropoietin (EPO) therapy within 2 months before the planned first dose of GX-E2 and Hb<10g/dL or No EPO therapy within a month (peritoneal dialysis) or 2 weeks (hemodialysis) before the planned first dose of GX-E2 and Hb<10g/dL.

Exclusion Criteria:

* Refractory to erythropoiesis stimulating agent (ESA) treatment
* History of blood transfusion within 3 months
* Donation or loss of blood for more than 400 milliliters (mL) within 8 weeks
* History of a known or suspected hypersensitivity, shock, or past history to the investigational drug or to similar ESA drugs
* Acute or chronic organ seizure disorder (including asthma and chronic obstructive pulmonary disease) which may be clinically deteriorated by the drug administration
* Active infection or history of infection that required intravenous injection of antibiotics in the last two months
* Grand Mal epilepsy
* Major surgery within 3 months other than access surgery
* Malignant tumor within 5 years other than successfully treated skin cancer that is not melanoma
* Ischemic stroke within 3 years
* Chest x-ray findings determined that they cannot participate in the study for clinically abnormal findings by the baseline chest x-ray findings or previously taken chest x-ray findings
* Uncontrolled hypertension
* Congestive heart failure more severe than NYHA functional class III; unstable Coronary artery disease (CAD); myocardial infraction within 3 months
* Uncontrolled arrhythmia
* High risk of thrombosis and embolism
* Systemic blood diseases (e.g. Pure red cell anemia, sickle cell anemia, myelodysplastic syndromes, hematologic malignancy, myeloma, hemolytic anemia)
* Absolute neutrophil count below 1,500 per microliter (uL) within screening periods
* Platelet count less than 5e10 per liter (L) within screening periods
* Hyperparathyrodism / hypothyrodism
* Splenomegaly caused by anemia or severe splenomegaly (>20cm)
* Blood aspartate aminotransferase/alanine aminotransferase (ALT/AST) concentration exceeds three times Upper Normal Limit of Normal (UNL)
* Blood total bilirubin concentration exceeds 1.5 times Upper Normal Limit of Normal (UNL)
* Blood albumin concentration below 3g per deciliter (dl)
* History of drug or alcohol abuse in the 6 months prior to the screening
* History of psychotropic or narcotic analgesic drugs dependence within 6 months prior to the screening
* Mental disorder or other central nervous system disorder determined that the study evaluation cannot be conducted
* Lack of understanding of the study and cooperation (one with no intention to give efforts to perform each evaluation visit and extend previously planned elective surgery)
* Female subjects with childbearing potential who are pregnant, breastfeeding or intends to become pregnant
* Participation in any drug study within 30 days prior to dosing
* Any other ineligible condition at the direction of the investigator that would be ineligible to participate the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
average change of Hemoglobin level | 6 weeks (Part A) & 14 weeks (Part B)
  change from baseline in Hemoglobin level

SECONDARY OUTCOMES:
change of red blood cell indices | 6 weeks (Part A) & 14 weeks (Part B)
  change from baseline in red blood cell indices
change of reticulocyte indices | 6 weeks (Part A) & 14 weeks (Part B)
  change from baseline in reticulocyte indices
incidence, degree, outcome of adverse event | 6 weeks (Part A) & 14 weeks (Part B)
  Incidence of adverse events
incidence, frequency, amount of blood transfusion | 6 weeks (Part A) & 14 weeks (Part B)
  Incidence of adverse events
immunogenicity: ratio of neutralizing antibody & binding antibody in subjects | 6 weeks (Part A) & 14 weeks (Part B)
  comparison from pre-treatment to post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Woo Yang, MD, Principal Investigator — 222 Banpo-daero, Seocho-gu, Seoul, Korea; Seok Joon Shin, MD, Principal Investigator — 56 Dongsuro, Pupyung-Gu, Incheon, Korea; Ki Young Na, MD, Principal Investigator — 82 Gumi-ro, 173 Beon-gil, Bundnag-gu, Seongnam-si, Gyeonggi-do, Korea; Ho cheol Song, MD, Principal Investigator — 327 sosaro, onemi-Gu, bucheon, Korea; Hyeong cheoon Park, MD, Principal Investigator — 211 Eonju-ro, Gangnam-gu, Seoul, Korea; Young Sun Kang, MD, Principal Investigator — 123 Jeokgeum-ro, Danwon-gu, Ansan-si, Gyeonggi-do, Korea; Eun Young Seong, MD, Principal Investigator — 176 Gudeok-ro, Seo-gu, Busan, Korea; Yong-Lim Kim, MD, Principal Investigator — 130 Dongdeok-ro, Jung-gu, Dae-gu, Korea; Sangho Lee, MD, Principal Investigator — 892 Dongnam-ro, Gangdong-gu, Seoul, Korea; Byung Chul Shin, MD, Principal Investigator — 365 Pilmun-daero, Dong-gu, Gwangju Metropolitan City; Su-Hyun Kim, MD, Principal Investigator — 102 Heukseok-ro, Dongjak-gu, Seoul, Korea; Hyung Wook Kim, MD, Principal Investigator — 93 Jungbu-daero, Paldal-gu, Suwon, Gyeonggi-do, Korea; Won Kim, MD, Principal Investigator — 20 Geonjiro Deokjin-gu, Jeonju-si, Jeollabuk-do, Korea; Young-il Jo, MD, Principal Investigator — 4-12 Hwayang-dong, Gwangjin-gu, Seoul, Korea; Sug Kyun Shin, MD, Principal Investigator — 100 Ilsan-ro, Ilsan-donggu, Goyang-si, Gyeonggi-do, Korea
Locations (5):
- South Korea (5):
  - Bucheon St. Mary's Hospital, Bucheon-si
  - Bundang Seoul National University College of Medicine, Gumi
  - The Catholic University of Korea Incheon St.Mary's Hospital, Incheon
  - Gangnam severance hospital, Seoul
  - Seoul St.Mary's Hospital, Seoul